CLINICAL TRIAL: NCT00534703
Title: Investigation of the Safety and Feasibility of AAV1/SERCA2a Gene Transfer in Patients With Chronic Heart Failure and a Left Ventricular Assist Device
Brief Title: Investigation of the Safety and Feasibility of AAV1/SERCA2a Gene Transfer in Patients With Chronic Heart Failure
Acronym: SERCA-LVAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination following Trial Steering Committee recommendation
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); Leducq Foundation (Other); Celladon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO782; 2007-002809-48 (EudraCT Number)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Chronic Heart Failure; Patients That Have Received a Left Ventricular Assist Device
Keywords: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAV1/SERCA2A (Active Comparator): SERCA gene therapy
  Interventions: Genetic: AAV1/SERCA2a
- Placebo (Placebo Comparator): Placebo (saline solution)
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: AAV1/SERCA2a — AAV1/SERCA2a will be delivered by a percutaneous method in the catheter laboratory. Dose: 1x 10^13 DRP (DNase resistant particles)
  Other Names: MYDICAR (R)
  Arms: AAV1/SERCA2A
Drug: Placebo — Placebo aliquots will be of the same composition as the investigational medicinal product with the absence of the active ingredient and will be visually indistinguishable from the medicinal product. Placebo is prepared and handled exactly as above in a blinded fashion.
  Arms: Placebo

SUMMARY:
The aim of the study is to determine the safety and feasibility of giving an adeno-associated viral vector expressing the sarcoplasmic reticulum calcium ATPase (SERCA2a), driven by the CMV promoter (AAV1-CMV-SERCA2a), to heart failure patients that have received a left ventricular assist device (LVAD) for an accepted clinical indication.

DETAILED DESCRIPTION:
It is a randomised, double-blind study of 24 patients that will be randomised to receive either the study drug (AAV1.SERCA2a) or placebo.

The purpose of gene transfer of SERCA2a is to improve systolic and diastolic function of the failing ventricle. Studies show that reduction of SERCA2a in failing ventricle is a key factor in depression of contraction, and that restoration of SERCA2a levels can improve function to near normal levels. The vector will be delivered during a cardiac catheterisation procedure by a 10-minute infusion into the coronary arteries.

Myocardial tissue is obtained at the time of LVAD placement, as a routine part of device implantation. Further samples will be obtained when the heart is transplanted or the LVAD removed. Measures of tissue inflammation as well as efficacy of gene transfer will be made by comparing these two samples. Recovery of contractile function of the heart will be assessed during attempts to wean patients from the LVAD using standard protocols.

The results will be assessed in conjunction with two companion studies which will start earlier in the US, one performing SERCA2a gene transfer with the same vector, but delivered by direct injection into the myocardium during LVAD insertion, and one using AAV1-CMV-SERCA2a delivered percutaneously in heart failure patients. The latter has both a dose-ranging and placebo-controlled arm.

ELIGIBILITY:
Inclusion criteria

* Patients that have had a left ventricular assist device (LVAD) implanted for chronic heart failure, where chronic heart failure is defined as at least 6 months
* Patients are clinically stable in the opinion of the clinical team looking after the patient
* Written informed consent

Exclusion criteria

* <18 or >70 years of age at the time of consent
* Pregnancy or within 6 months of giving birth
* Women of child-bearing potential not using an effective method of contraception
* Men not using an effective method of contraception
* Suspected or active viral, fungal or parasitic infection within 48 hours prior to administration of IMP, in the opinion of the investigator*.
* Patients at a high risk of thrombosis in the opinion of the investigator
* Patients with a previous episode of LVAD thrombosis
* Patients with persistently raised lactate dehydrogenase (LDH >2.5 ULN)
* Patients requiring triple anticoagulation i.e. warfarin and dual anti-platelet
* Patients participating in another clinical trial
* Patients unable to comply with the protocol mandated procedures for social or other reasons, in the opinion of the investigator and primary care physician

  * Eligible, enrolled and randomised patients who develop an infection will have study treatment delayed until 7 or more days after the time point when infection is no longer clinically evident.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sian Harding, Principal Investigator — Imperial College London; Alexander Lyon, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - Harefield Hospital, Royal Brompton and Harefiled NHS Trust, Middlesex

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AAV1/SERCA2A | Placebo
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAV1/SERCA2A | Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Continuous [Mean (Full Range); unit: years] | 41 [29 to 69] | 49 [49 to 49] | 42.6 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 0 | 4
  Black | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety and Feasibility of Administering AAV1/SERCA2a to LVAD Patients
Description: Safety is defined as the incidence of patients experiencing death and major adverse cardiovascular events, and out of range laboratory values. Both AAV1/SERCA2a treated cohorts (NAb+ and NAb-) will be compared to the placebo group.
Time Frame: 6 months
Population: The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and results have been presented taking a descriptive approach instead
Measure: Count of Participants; unit: Participants
Groups:
- AAV1/SERCA2A: SERCA gene therapy
  AAV1/SERCA2a: AAV1/SERCA2a will be delivered by a percutaneous method in the catheter laboratory. Dose: 1x 10^13 DRP (DNase resistant particles)
  No statistical analyses have been specified for this primary end point. It is expected there is at least one statistical analysis for each primary end point.
  Justification: The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety.
- Placebo: Placebo (saline solution)
  Placebo: Placebo aliquots will be of the same composition as the investigational medicinal product with the absence of the active ingredient and will be visually indistinguishable from the medicinal product. Placebo is prepared and handled exactly as above in a blinded fashion.
  No statistical analyses have been specified for this primary end point. It is expected there is at least one statistical analysis for each primary end point.
  Justification: The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety.
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 4 | 1
Participants | NA — The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety. | NA — The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety.

2. Secondary Outcome: Number of Participants With Exogenous Viral Vector Genome in the Myocardium Measured by qPCR for the Viral DNA
Description: The trial was terminated early with only 5 subjects enrolled. As a result full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 4 | 1
Participants | 0 | 0

3. Secondary Outcome: Left Ventricular Function (LVEF)
Description: Left ventricular function assessed by echocardiography and exercise capacity (6MWT, MVO2) during minimal LVAD support (low/no flow settings depending upon device) LVEF expressed as %
Time Frame: 6 months
Population: Note: The trial was terminated early with only 5 subjects enrolled. As a result, full statistical analysis for both primary and secondary outcomes was impossible and results have been presented using a descriptive approach
Measure: Count of Participants; unit: Participants
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 4 | 1
Participants | NA — Note: The trial was terminated early with only 5 subjects enrolled. As a result, full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety. | NA — Note: The trial was terminated early with only 5 subjects enrolled. As a result, full statistical analysis for both primary and secondary outcomes was impossible and a more pragmatic approach was undertaken to assess product safety.

4. Secondary Outcome: Levels of SERCA2a Protein
Time Frame: 6 months
Population: Data not collected due to early termination of the trial
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Other Relevant Proteins e.g. Phospholamban, the Sarcoplasmic Reticulum Calcium Release Channel, the Na+/Ca2+-Exchanger.
Time Frame: 6 months
Population: Data not collected due to early termination of the trial
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Function of Isolated Myocytes
Time Frame: 6 months
Population: Data not collected due to early termination of the trial
Arm/Group | AAV1/SERCA2A | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | AAV1/SERCA2A | Placebo
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAV1/SERCA2A (N=4) | Placebo (N=1)
LVAD Alarm (Product Issues) | 1 (1) | 0 (0) — LVAD Alarm and power increase with hospital admission
Worsening heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Heart transplantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAV1/SERCA2A (N=4) | Placebo (N=1)
Vessel puncture, site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Iron deficiency - Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Site Bleeding (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Device Alarm Issue (Product Issues) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes